CLINICAL TRIAL: NCT04409730
Title: Reliability of Photographic Posture Analysis in Children With Cerebral Palsy and Its Relationship With Trunk Control and Motor Functions
Brief Title: Photographic Posture Analysis in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Pt, PhD, Associate Professor, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: KA19/126
Record Dates: First submitted 2020-05-22; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Posture Disorders in Children; Cerebral Palsy
Keywords: trunk; posture analysis; cerebral palsy; performance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with Cerebral Palsy (Experimental): Aged 5-12 years, diagnosed as spastic diplegia or hemiplegia , having a level of "I, II, III" according to GMFCS
  Interventions: Other: Photographic Posture Analysis

INTERVENTIONS:
Other: Photographic Posture Analysis — Postural evaluation was done using the photographic method. All measurements were made by two researchers experienced in postural analysis evaluation. Canon camera and national geographic tripod with double spirit level were used for evaluation. The camera was placed on a 115 cm high tripod, 1.5 m away from the subjects. Spirit levels have been adjusted so that the tripod is completely flat on the ground. The tripod was taped to the floor to maintain the same distance between the camera and the participants. Six photographs of each child whose feet on the ground, in a free-sitting position, 3 from the front and 3 sides were taken by the researchers.

SUMMARY:
Cerebral palsy (CP), which is the largest group of patients among pediatric neuromuscular diseases, is a non-progressive permanent disorder that affects muscle control, movement, posture and balance. The purpose of this study; to evaluate the reliability of photographic posture analysis in the sitting position in children with CP and to examine the relationship between the results of photographic posture analysis with the motor performances and trunk control of children with CP.Children with CP were included in the study according to the following criteria; aged 5-12 years, diagnosed as spastic diplegia or hemiplegia , having a level of "I, II, III" according to GMFCS. Postural evaluation was done using the photographic method. Trunk control was evaluated with Trunk Control Measurement Scale,Motor performance of children was evaluated with Gross Motor Function Measure-88. ICC values for photographic posture analysis was found to be highly reliable.

DETAILED DESCRIPTION:
Sitting position is of great importance in the development of upper extremity functions, orthogonal functional skills, personal care, cognitive, perceptual and social skills in children with cerebral palsy and these kids spend most of their time in a sitting position.There are goniometer, inclinometer, flexicurve, spinal mouse, and modified head posture spinal curvature ınstrument tools for posture analysis in the sitting position.However, none of these measurement tools have been validated for validity and reliability studies of head and trunk posture measurement in the sitting position in children with CP. Methods such as magnetic resonance (MR) and x-ray used in posture evaluation provide clear images of reference points and are the gold standard in the literature. However, they are not preferred much because they are expensive and contain radiation.Photographic posture analysis can be considered as a measurement method such as posture analysis methods using the gravity line. It is a digital, more objective measurement method that measures linear distances and angles using anatomical reference points using specially designed software. Clinical use of photographic posture analysis is recommended in the literature, as it is an accurate and objective method, preventing radiation exposure.The purpose of this study; to evaluate the reliability of photographic posture analysis in the sitting position in children with CP and to examine the relationship between the results of photographic posture analysis with the motor performances and trunk control of children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-12 years,
* Diagnosed as spastic diplegia or hemiplegia,
* Having a level of "I, II, III" according to GMFCS

Exclusion Criteria:

* Children who could not cooperate,
* Have undergone spinal surgery, had botulinum toxin (BoNT) and surgical treatment in the last 6 months
* Had another neurodevelopmental or congenital disease other than CP

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Photographic Posture Analysis | 45-60 minutes
  Postural evaluation was done using the photographic method. All measurements were made by two researchers experienced in postural analysis evaluation. Canon camera and national geographic tripod with double spirit level were used for evaluation Six photographs of each child whose feet on the ground, in a free-sitting position, 3 from the front and 3 sides were taken by the researchers

SECONDARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | 30-40 minutes
  Trunk control was evaluated with Trunk Control Measurement Scale is a scale that measures the static and dynamic sitting balance in children with CP. It consists of 15 items in total, 1-5 items measure Static Sitting Balance, 6-15 items measure dynamic sitting balance. Static sitting balance assesses the ability of children to maintain the trunk posture as they move their upper and lower limbs in the sitting posture. Dynamic sitting balance is divided into two sub-scales; selective motion control scale and dynamic reach scale. The maximum score that can be obtained from the test is 58. Higher scores perform better.
Gross Motor Function Measure-88 (GMFM-88) | 30-45 minutes
  GMFM-88 is a standardized observational test designed to measure the motor development levels of children with SP and their changes over time. It consists of five main headings and 88 items: lying and rolling; sitting; crawling and kneeling; standing; walking, running, and jumping. 17 of the 88 items are on the lying and rolling part, 20 on the sitting part, 14 on the crawling and kneeling part, 13 on the standing part, and 24 on the walking, running, and jumping part. Likert scale is used in scoring. The child gets 0 points if he / she cannot start the movement, 1 if he / she can start the movement independently, 2 if he / she can partially complete the movement, and 3 if he / she can complete the movement independently. A 5-year-old child with normal development is expected to score full of 88 items. The GMFM-88 was administered to the children by therapists trained in its use and tested to ensure an adequate level of competence by using a criterion test videotape

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Çömük Balcı, Pt,PhD, Study Director — Baskent University
Locations (1):
- Baskent University, Ankara, Etimesgut, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No